CLINICAL TRIAL: NCT07009587
Title: Ionizing Radiation During Endoscopic Procedures: a Single-center, Prospective Study of Dose Reference Levels.
Brief Title: Ionizing Radiation During Endoscopic Procedures (ENDORAY Study)
Acronym: ENDORAY
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-06-010
Record Dates: First submitted 2025-05-16; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Gastro-Intestinal Disorder
MeSH Terms: conditions — Digestive System Diseases | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopy
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — endoscopic procedure

SUMMARY:
The primary objective of this prospective study was to describe the evolution of dose reference levels (DRLs) in a specialized French center during endoscopic procedures involving ionizing radiation and performed without a radiology technician. The secondary objective was to assess the influence of the operator on the recorded dose for each procedure.

DETAILED DESCRIPTION:
This prospective study, approved by the Institutional Review Board (IRB) of the Groupement de Coopération Sanitaire Ramsay Santé (approval no. 2019-06-010), was conducted in the endoscopy unit of Jean Mermoz Hospital (Lyon, France).

To standardize practices, all operators underwent blended training (3 hours of e-learning and 3 hours of hands-on training on the Shine Enhancer system), which was completed and validated on June 25, 2018. As per guidelines, the graphic (cine) mode was never used. Only the latest fluoroscopic images were printed and archived.

The database includes all consecutive patients who underwent an endoscopic procedure between June 26, 2018, and December 31, 2021. Each report was retrospectively reviewed to confirm the therapeutic intention (intention-to-treat).

Initially, only the type of procedure and the dose-area product (DAP) were recorded. From October 7, 2019, fluoroscopy time (FT) was also systematically collected.

Six experienced endoscopists performed all procedures. The patient's position varied depending on the procedure, although most were performed in the supine position under general anesthesia. No radiologic technician was present during the procedures. The fluoroscopic system was entirely managed by the endoscopist, including all parameter adjustments (distance between patient and detector, use of pulsed vs continuous fluoroscopy, collimation, duration, etc.).

Two mobile C-arm X-ray systems were used throughout the study: Siemens Arcadis and GE OEC Fluorostar, both under-couch systems.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, who have been informed of the research;
* Patients who have undergone an endoscopic procedure under radiological control
* Subjects for whom all data concerning the methods of exposure to ionizing radiation are available;

Exclusion Criteria:

* Patient under legal protection, guardianship, or curatorship;
* Patient who has indicated their opposition to the use of their medical data (by completing and returning the opposition form that will be sent to them).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients participating in the study underwent a digestive endoscopy under radiological control.
Sampling Method: Non-Probability Sample
Enrollment: 2782 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
dose reference level | Periprocedural
  Assessment of dose reference levels (DRLs) with the Dose Area Product (DAP) collected for each procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No